CLINICAL TRIAL: NCT02157181
Title: Study on the Treatment of Hairy Cell Leukaemia Variant and Relapsing Hairy Cell Leukaemia
Brief Title: Treatment of Hairy Cell Leukaemia Variant and Relapsing Hairy Cell Leukaemia With Cladribine Plus Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jurgen Barth (Other)
Responsible Party: Sponsor-Investigator, Jurgen Barth, Professor Dr. med Mathias Rummel, University of Giessen
Organization: University of Giessen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL 4-2004
Record Dates: First submitted 2014-05-21; First posted 2014-06-05 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hairy Cell Leukemia (HCL)
Keywords: HCL variant; HCL relapse; Risk stratified
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Cladribine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCL, 2CdA +/- Rituximab (Experimental): Risk stratification
  1. HCL variant will be treated with cladribine plus rituximab, independent of previous therapy
  2. Relapses of HCL will be treated with cladribine plus rituximab, duration of remission of the previous therapy is < 3 years.
  3. All repeated relapses (> 1st relapse) after previous therapies with purine analogues and/or interferon will be treated with cladribine plus rituximab.
     Cladribine (LITAK®) 0.14 mg/kg daily Days 8-12 subcutaneous bolus injection Rituximab (Mabthera®) 375 mg/m2 daily Days 1, 8, 15, 22 infusion
  4. Relapses of HCL will be treated with cladribine monotherapy, if the duration of remission of the previous therapy is > 3 years.
  Cladribine (LITAK®) 0.14 mg/kg daily Days 1-5 subcutaneous bolus injection
  Interventions: Drug: 2CdA +/- Rituximab

INTERVENTIONS:
Drug: 2CdA +/- Rituximab — Cladribine 0.14 mg/kg daily subcutaneous bolus injection Rituximab 375 mg/m² infusion
  Other Names: Cladribine, Syn 2CdA, (LITAK®) 0.14 mg/kg; Rituximab (Mabthera®; Rituxan®) 375 mg/m²

SUMMARY:
The study will test the effectiveness (rate of complete remissions, total remission rate and duration of remission) and toxicity of the combined immuno/chemotherapy with subcutaneous cladribine (LITAK®) plus anti-CD20* antibody rituximab in patients requiring treatment for relapsed hairy cell leukaemia or hairy cell leukaemia variant independent of any previous therapy.

CD20* = cluster of differentiation antigen 20

DETAILED DESCRIPTION:
The trial is a prospective, multi-centre, open Phase II study on patients with hairy cell leukaemia variant or with relapsed hairy cell leukaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified hairy cell leukaemia (HCL) Hairy cell leukaemia variant (HCLv) or
* Relapse of hairy cell leukaemia after therapy with cladribine or pentostatin
* Need for treatment is indicated (see 4.3 below)
* Age at least 18 years
* General state of health according to WHO 0-2
* Written declaration of consent by the patient
* Current histology, which should not be older than 6 months, is necessary

Exclusion Criteria:

* Patients, who do not fulfil the above-mentioned inclusion criteria.
* Patients with severe functional limitations of the heart according to New York Heart Association III / IV, of the lung according to WHO degree III / IV, the liver (bilirubin > 2mg/dl, alkaline phosphatase, raised GOT and GPT (glutamate- pyruvate transaminase) values more than twice normal), diseases of the central nervous system, including psychoses. Creatinine > 2 mg/dl, or creatinine clearance < 50 mg/min
* Patients with proven HIV infections
* Patients with active hepatitis
* Patients with other florid infections
* Patients with anamnesis / diagnosis of another malignant disease (other than nonmelanoma associated skin tumours or stage 0 in situ carcinoma of the cervix)
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-06; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of complete remissions (CR) | 4 months after treatment
  Determination of the rate of complete remission and duration of remission after one cycle of subcutaneous cladribine (LITAK®) plus four administrations of rituximab
  * in patients with hairy cell leukaemia variant
  * in patients with relapsed hairy cell leukaemia

SECONDARY OUTCOMES:
Overall remission rate (ORR) | 4 months after treatment
  The rate of CR + PR will be determined

OTHER OUTCOMES:
Acute and late toxicity | From day 1 of treatment period up to 120 months
  All kind of adverse events, laboratory abnormalities, infections, unplanned hospitalisations will be measured
Degree of induced immunodeficiency | From day 1 of treatment period up to 120 months
  Degree of immunosupression with CD4/CD8 quotient as indicating biomarker will be measured.
  Duration of immunosupression as well as infectious and other complications which result from therapy will be reported
Frequency of secondary neoplasia during the life-long follow-up period | From day 1 of treatment period up to 120 months
  Rate of secondary neoplasia as safety issue will be determined
Overall survival (OS) | From achieving a remission until death
  Determination of the overall survival times of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Mathias J Rummel, Prof. Dr., Principal Investigator — Justus-Liebig-University | University Hospital | Medicinal Clinic IV
Locations (46):
- Germany (46):
  - Community based hemato-oncology medical office, Ansbach
  - Community based hemato-oncology medical office, Aschaffenburg
  - Community based hemato-oncology medical office, Celle
  - St.-Johannes-Hospital, Dortmund
  - Städtische Kliniken Esslingen, Esslingen am Neckar
  - Universitätsklinik Frankfurt, Frankfurt am Main
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Community based hemato-oncology medical office, Fürth
  - University Clinic | Med. Cinic IV Justus-Liebig-University, Giessen
  - Wilhelm-Anton-Hospital, Goch
  - Kath. Krankenhaus Hagen gem. GmbH, Hagen
  - Community based hemato-oncology medical office, Halle
  - Community based hemato-oncology medical office, Hamburg
  - Meditinische Hochschule (MHH), Hanover
  - Community based hemato-oncology medical office, Heidelberg
  - Marienhospital Herne/ Klinikum der Ruhr-Universität Bochum, Herne
  - Community based hemato-oncology medical office, Hilden
  - Community based hemato-oncology medical office, Hildesheim
  - Klinikum Idar-Oberstein, Idar-Oberstein
  - Community based hemato-oncology medical office, Jena
  - Community based hemato-oncology medical office, Kassel
  - Community based hemato-oncology medical office, Kiel
  - Community based hemato-oncology medical office, Koblenz
  - Community based hemato-oncology medical office, Kronach
  - Community based hemato-oncology medical office, Leer
  - Community based hemato-oncology medical office, Leipzig
  - Städtische Kliniken, Leverkusen
  - Community based hemato-oncology medical office, Magdeburg
  - Community based hemato-oncology medical office, Marburg
  - Klinik Schwäbisch Gmünd / Staufer Klinik, Mutlangen
  - Community based hemato-oncology medical office, München
  - Klinikum Großhadern, München
  - Community based hemato-oncology medical office, Neunkirchen
  - Community based hemato-oncology medical office, Neuwied
  - Community based hemato-oncology medical office, Niddatal
  - Community based hemato-oncology medical office, Nuremberg
  - MVZ Klinikum Osnabrück, Osnabrück
  - Community based hemato-oncology medical office, Pforzheim
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - St. Josefs-Krankenhaus, Potsdam
  - Community based hemato-oncology medical office, Schweinfurt
  - St. Marien-Krankenhaus, Siegen
  - Community based hemato-oncology medical office, Straubing
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Community based hemato-oncology medical office, Villingen
  - Community based hemato-oncology medical office, Wolfsburg